CLINICAL TRIAL: NCT00039559
Title: Ovarian Cancer Screening Pilot Trial in High Risk Women
Brief Title: Clinical Trial to Screen Participants Who Are at High Genetic Risk for Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Skates, Steven Skates PhD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDR0000069397; MGH-000084; NCT00301743 (obsolete NCT alias)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Ovarian Cancer
Keywords: ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Early detection (Other)
  Interventions: Other: Early detection

INTERVENTIONS:
Other: Early detection — CA125 is measured in blood and the longitudinal results interpreted with a statistical algorithm to determine if there has been a significant increase from baseline.

SUMMARY:
RATIONALE: Screening tests may help doctors detect cancer cells early and plan more effective treatment for ovarian cancer.

PURPOSE: Screening trial to determine the significance of cancer antigen 125 (CA125) levels in detecting ovarian cancer in participants who have a high genetic risk of developing ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of prospective ovarian cancer screening studies within the Cancer Genetics Network and other NCI ovarian programs for participants who are at high genetic risk for developing ovarian cancer.
* Identify the logistical issues of screening these participants and their solutions within this framework.
* Establish normal ranges and distributions of CA125 values over time within and between high-risk participants, with subclassification by pre- or post-menopausal status, estrogen-replacement therapy usage, and prior prophylactic oophorectomy.
* Estimate the specificity and positive predictive value of the "risk of ovarian cancer algorithm" (ROCA) suitable for designing a definitive trial of screening for ovarian cancer in high-risk participants.
* Establish a longitudinal serum and plasma biorepository for retrospective evaluation of other promising biomarkers with special relevance to inherited ovarian and breast cancer risk.

OUTLINE: This is a multicenter study. Participants with 1 or 2 ovaries are assigned to group A, whereas participants with prior prophylactic bilateral oophorectomy are assigned to group B (closed to accrual as of 10/18/04).

At baseline, participants who are not eligible by breast cancer susceptibility gene (BRCA) mutation criteria or family history criteria undergo a probability of having a BRCA mutation given family history of cancer (BRCAPRO) evaluation. Participants in both groups complete a questionnaire requesting demographic information and a personal and family health history at baseline and a questionnaire requesting hospitalization or cancer diagnosis information after each blood test. Participants in both groups also complete health status questionnaires once every 3 months for 6 months-7 years. Participants undergo blood draws for measurement of CA125 levels once every 3 months for 6 months-7 years. For each CA125 measurement, the risk of ovarian cancer algorithm (ROCA) is calculated.

Group A (1 or 2 ovaries at baseline):

* Participants are assigned to 1 of 2 subgroups based on ROCA.

  * Subgroup A1: Participants with normal-risk for ovarian cancer (ROCA less than 1%) continue CA125 screening as above.
  * Subgroup A2: Participants with intermediate-risk for ovarian cancer (ROCA more than 1% but less than 10%) or elevated-risk for ovarian cancer (ROCA more than 10%) undergo transvaginal sonography (TVS). Participants with elevated-risk undergo an additional blood draw for a confirmatory CA125 level prior to TVS. Participants with normal TVS continue CA125 screening as above. Participants with abnormal TVS are referred to a gynecologic oncologist who decides whether standard clinical intervention for potential ovarian cancer is needed. Participants who are not referred for standard clinical intervention continue CA125 screening as above. Participants who are referred for standard clinical intervention, have at least 1 ovary remaining, and are found to have no malignancy continue CA125 screening as above. Participants who are referred for standard clinical intervention, are found to have no malignancy, and then undergo prophylactic bilateral oophorectomy proceed to CA125 screening as in group B below. Participants who are referred for standard clinical intervention and are found to have malignancy are taken off study.

Group B (no ovaries at baseline) (closed to accrual as of 10/18/04):

* Participants are assigned to 1 of 2 subgroups based on ROCA.

  * Subgroup B1: Participants with normal-risk for ovarian cancer (ROCA less than 5%) continue CA 125 screening as above.
  * Subgroup B2: Participants with elevated-risk for ovarian cancer (ROCA more than 5%) undergo an additional blood draw for a confirmatory CA125 level and are then referred to a gynecologic oncologist who decides whether standard clinical intervention for potential ovarian cancer is needed. Participants who are not referred for standard clinical intervention continue CA125 screening as above. Participants who are referred for standard clinical intervention and are not found to have malignancy continue CA125 screening as above. Participants who are referred for standard clinical intervention and are found to have malignancy are taken off study.

Patients are followed for clinical diagnosis for 1 additional year.

PROJECTED ACCRUAL: Approximately 2,430 participants will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Participant meet the criteria for one of the following conditions:

  * Participant has tested positive for a mutation in the breast cancer susceptibility gene 1 (BRCA1) or breast cancer susceptibility gene 2 (BRCA2) or has a first- or second-degree relative with a BRCA1 or BRCA2 mutation
  * At least 2 ovarian or breast cancers (including ductal carcinoma in situ) have occurred among the participant and her first- and second-degree relatives within the same lineage

    * Condition may be satisfied by multiple primary cancers in the same person
    * Where breast cancer is required to meet this criterion, at least 1 breast cancer patient must have been pre-menopausal (age 50 and under at diagnosis if age at menopause unknown)
  * Participant is of Ashkenazi Jewish ethnicity and either has had breast cancer or has 1 first-degree or 2 second-degree relatives with breast cancer (including ductal carcinoma in situ) or ovarian cancer

    * Where breast cancer is required to meet this criterion, at least 1 breast cancer patient must have been pre-menopausal (age 50 and under at diagnosis if age at menopause unknown)
  * Probability of carrying a BRCA1 or BRCA2 mutation exceeds 20% as calculated by BRCAPRO, given family pedigree of breast cancer (including ductal carcinoma in situ) and ovarian cancer
* Participant must have no prior or concurrent ovarian cancer (including low malignant potential (LMP) cancers) or primary papillary serous carcinoma of the peritoneum
* Participant must not be negative for the same BRCA1 or BRCA2 mutation for which a first- or second-degree relative has tested positive
* Participants who test negative for BRCA1 or BRCA2 mutation are still eligible if the pedigree or BRCAPRO criteria are satisfied, including Ashkenazi women who test negative for the three founder mutations
* Documentation of family history is by participant's self-report
* In relatives, ovarian cancer is defined as invasive ovarian epithelial cancers, fallopian tube cancers, or primary papillary serous carcinoma of the peritoneum
* Germ cell or granulosa tumors or LMP ovarian cancers do not qualify
* First- and second-degree relatives include half siblings of the participant or her first-degree relative

PATIENT CHARACTERISTICS:

Age:

* 30 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* No hemophilia or other bleeding disorders
* No serious anemia

Hepatic:

* Not specified

Renal:

* Not specified

Pulmonary:

* No emphysema

Other:

* Not pregnant
* Fertile patients must use effective contraception
* No psychiatric, psychological, or other conditions that would preclude informed consent
* No concurrent untreated malignancy except nonmelanoma skin cancer
* No medical conditions that would preclude blood draws during study
* No chronic infectious disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 months since prior adjuvant anticancer chemotherapy

Endocrine therapy:

* Prior or concurrent adjuvant hormonal therapies (e.g., tamoxifen, leuprolide, or goserelin) allowed
* Concurrent hormonal therapies (e.g., tamoxifen) for prevention allowed

Radiotherapy:

* At least 3 months since prior adjuvant anticancer radiotherapy

Surgery:

* At least 3 months since prior intraperitoneal surgery (laparoscopy or laparotomy)
* No prior prophylactic oophorectomy

Other:

* At least 5 years since prior non-hormonal treatment for metastatic malignancy
* No concurrent participation in other ovarian cancer early detection trials

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2430 (Estimated)
Dates: Start 2002-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of early detection for ovarian cancer | Up to one year since last blood test

SECONDARY OUTCOMES:
Specificity of early detection | Up to one year from last blood test

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Skates, PhD, Study Chair — Massachusetts General Hospital
Locations (1):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States